CLINICAL TRIAL: NCT06277310
Title: Personalized End of Life Care in Safety-Net Hospitals: Implementation of the 3 Wishes Project
Brief Title: Wishes to Improve Support and Humanity at End-of-life in Safety-net Hospitals
Acronym: WISHES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Olive View-UCLA Education & Research Institute (Other); LAC+USC Medical Center (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Thanh H. Neville, MD, MSHS, Associate Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 3WP in SNH; 5R01NR020773 (NIH)
Record Dates: First submitted 2024-02-13; First posted 2024-02-26 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: End of Life
MeSH Terms: conditions — Death

STUDY DESIGN:
Intervention Model Description: This is a before and after stepped wedge study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 3WP intervention (Experimental): families of patients whose loved ones died in the ICU where the 3 Wishes Program has been implemented
  Interventions: Other: 3 Wishes Project

INTERVENTIONS:
Other: 3 Wishes Project — palliative care initiative in which clinicians elicits and implements small acts of kindness for dying patients and their families

SUMMARY:
Dignified and compassionate end-of-life (EOL) care is a cornerstone of high-quality, patient-centered care, but in safety-net hospitals EOL care is often overlooked, considered too late, or not at all. By eliciting and implementing final wishes for dying patients, the 3 Wishes Project (3WP) has demonstrated, in tertiary academic centers, that acts of compassion can improve the EOL experience and help families cope with loss. The investigators propose to implement the 3WP in safety-net hospitals where there are less resources and more diverse, disadvantaged patient populations, and hypothesize that there will be similar positive effects on the EOL experience for patients, families, and clinicians.

DETAILED DESCRIPTION:
Compassionate end-of-life (EOL) care is foundational to medicine, but providing patients and families in safety-net hospitals (SNHs) with the sense that they are physically and emotionally supported during a patient's terminal hospitalization can be challenging. SNHs are public hospitals that primarily provide services to low-income and uninsured patients on a minimal budget. Although high quality EOL care is an important unmet need in SNHs, its provision is fraught with barriers and challenges. Language barriers, low health literacy, and cultural differences can make it difficult for families in SNHs to perceive empathy and support during the EOL. Deaths in the intensive care unit (ICU) for underserved families can be traumatic, and families of patients who die in the ICU often suffer from depression and post-traumatic stress disorder. Palliative care interventions are needed, but implementation is often resource-prohibitive.

The 3 Wishes Project (3WP) is a palliative care intervention that aims to achieve a dignified and compassionate EOL experience by empowering the clinical team to elicit and fulfill small wishes for critically ill patients who are dying in the ICU. Although the 3WP has been shown to improve a family's experience of their loved one's EOL care, ease bereavement, and enhance clinician work satisfaction in academic centers, it has not been implemented and evaluated in low-resource hospitals. The investigators believe that this patient-centered and clinician-partnered initiative can improve the EOL experience in SNHs, but that it must be adapted to the contextual differences and needs of low-resource hospitals.

Investigators propose to obtain and use stakeholder input to customize a multi-component 3WP Toolkit that will facilitate 3WP implementation in SNHs. Using the tailored Toolkit, the investigators will implement and evaluate the 3WP in the three SNHs of the Los Angeles County Department of Health Services. The investigators will conduct a pragmatic type 2 hybrid effectiveness-implementation study to evaluate the quality of EOL ICU care, bereaved families' psychological symptoms, and clinician burnout as compared to usual care. The Consolidated Framework for Implementation Research (CFIR) and the RE-AIM (Reach, Effectiveness, Adoption, Implementation, and Maintenance) framework will be used to guide a mixed-methods evaluation of the 3WP implementation in SNHs.

ELIGIBILITY:
Inclusion Criteria:

* For participation in the 3WP, if there was a decision to withdraw life support or the health care team agreed that the patient's probability of dying in the hospital or on discharge to hospice was >95% For surveys, next of kin/surrogate of a patient who died in the ICU during the study period For surveys, speaks English or Spanish

Exclusion Criteria:

* <18 years old
* does not speak english or spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Families' assessment of the quality of end-of-life, particularly in emotional and spiritual support. | 3 months after patient's death (families will be surveyed 3 months after the date of death).
  Bereaved families of patients who died in the ICU will complete an after-death survey, which includes the Bereaved Family Survey (BFS). The BFS asks questions regarding the family's perception of the patient's end of life care. We will also use a question from the FS-ICU (family satisfaction with ICU) to assess whether family felt supported in final hours of patient's life.

SECONDARY OUTCOMES:
Family anxiety and depression | 3 months after patient's death (families will be surveyed 3 months after the date of death).
  The Hospital Anxiety and Depression scale (HADS) will part of the after death survey.
Nurse Burnout | 6 months and 1 year after
  Nurses will be asked to complete a survey (MBI) that evaluates nursing burnout before and after 3WP implementation.
Family PTSD | 3 months after patient's death (families will be surveyed 3 months after the date of death).
  The PTSD Checklist for DSM-V (PCL-5) is part of the after death survey

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - LA General Hospital, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Olive View Medical Center, Sylmar, California
  - Harbor-UCLA, Torrance, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neville TH, Clarke F, Takaoka A, Sadik M, Vanstone M, Phung P, Hjelmhaug K, Hainje J, Smith OM, LeBlanc A, Hoad N, Tam B, Reeve B, Cook DJ. Keepsakes at the End of Life. J Pain Symptom Manage. 2020 Nov;60(5):941-947. doi: 10.1016/j.jpainsymman.2020.06.011. Epub 2020 Jun 21. PMID 32574658
- [Background] Vanstone M, Neville TH, Clarke FJ, Swinton M, Sadik M, Takaoka A, Smith O, Baker AJ, LeBlanc A, Foster D, Dhingra V, Phung P, Xu XS, Kao Y, Heels-Ansdell D, Tam B, Toledo F, Boyle A, Cook DJ. Compassionate End-of-Life Care: Mixed-Methods Multisite Evaluation of the 3 Wishes Project. Ann Intern Med. 2020 Jan 7;172(1):1-11. doi: 10.7326/M19-2438. Epub 2019 Nov 12. PMID 31711111
- [Background] Vanstone M, Neville TH, Swinton ME, Sadik M, Clarke FJ, LeBlanc A, Tam B, Takaoka A, Hoad N, Hancock J, McMullen S, Reeve B, Dechert W, Smith OM, Sandhu G, Lockington J, Cook DJ. Expanding the 3 Wishes Project for compassionate end-of-life care: a qualitative evaluation of local adaptations. BMC Palliat Care. 2020 Jun 30;19(1):93. doi: 10.1186/s12904-020-00601-5. PMID 32605623
- [Background] Cook DJ, Clarke FJ, Neville TH, Hoad N, Boyle A, Woods A, Dionne JC, Dennis BB, Toledo F, Tam B, Swinton M, Reid J, Vanstone M. The 3 Wishes Project: toward spiritual care at the end of life. Pol Arch Intern Med. 2023 Mar 29;133(3):16465. doi: 10.20452/pamw.16465. Epub 2023 Mar 29. No abstract available. PMID 36994496
- [Background] Neville TH, Taich Z, Walling AM, Bear D, Cook DJ, Tseng CH, Wenger NS. The 3 Wishes Program Improves Families' Experience of Emotional and Spiritual Support at the End of Life. J Gen Intern Med. 2023 Jan;38(1):115-121. doi: 10.1007/s11606-022-07638-7. Epub 2022 May 17. PMID 35581456
- [Derived] Neville TH, Walling A, Wenger NS, Mittman BS, Tseng CH, Chang D, Cook D, Marentes Ruiz CJ, Cassano H, Beers E, Gadgil R, Kamangar N, Blake N, Tarn DM. Implementation and evaluation of the 3 Wishes Project in safety-net hospitals: Protocol for a hybrid effectiveness-implementation study. PLoS One. 2025 May 2;20(5):e0320843. doi: 10.1371/journal.pone.0320843. eCollection 2025. PMID 40315279